CLINICAL TRIAL: NCT00118677
Title: Long-Term Supervised Treatment Interruption in HIV-Infected Patients Who Started Antiretroviral Treatment With CD4 Over 350/mm3 and Plasma HIV RNA Below 50 000/mL ANRS 116 Trial SALTO
Brief Title: Long-Term Supervised Treatment Interruption in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 116 SALTO
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

INTERVENTIONS:
Procedure: Treatment interruption

SUMMARY:
This trial is aimed at studying the safety of long term supervised treatment interruption in HIV infected patients with CD4 over 350/mm3 and plasma HIV RNA under 50 000/mL. Another aim of this study is to assess the immunological and virological factors associated with the duration of treatment interruption.

DETAILED DESCRIPTION:
The limitations of the drugs used against HIV include their toxicity, their tolerability, their propensity to induce resistance when not taken with absolute regularity and their cost. Treatment interruption in patients receiving antiretroviral treatment in the setting of chronic infection are associated with viral rebound and rapid CD4 T cell decrease conducting to antiretroviral therapy restart.

In patients with high CD4+ cell counts (patients receiving treatment of chronic infection with controlled viremia and patients who are receiving HAART now in whom treatment would not have been started based on current guidelines), we evaluated the safety of long term supervised treatment interruption. Another aim of this study was to assess the immunological and virological factors associated with the duration of treatment interruption (proviral HIV DNA at baseline and during follow-up, plasma HIV RNA at baseline and during follow-up, CD4 T cell and CD8 T cell HIV specific responses at baseline and after 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Males and non pregnant females
* 18 years of age and older
* Who have confirmed laboratory diagnosis of HIV infection
* Started on first line antiretroviral treatment with CD4 over 350/mm3 and plasma HIV RNA below 50 000/mL
* Ongoing Antiretroviral therapy at inclusion with CD4 over 450/mm3 and plasma HIV RNA below 5000/mL

Exclusion Criteria:

* HBV-HIV co-infection receiving lamivudine therapy
* Ongoing immunotherapy including IL2, interferon or HIV specific vaccine
* Pregnancy or project of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who did not resume antiretroviral treatment at 12 months

SECONDARY OUTCOMES:
Time to resume antiretroviral treatment with CD4 cell count equal or below 300/mm3
Proportion of patients who did not resume antiretroviral treatment at M 24 and M 36
Predictive factors associated with the time of restart of antiretroviral therapy: Proviral HIV DNA at baseline and during follow-up
Plasma HIV RNA at baseline and during follow-up
CD4 T cell and CD8 T cell HIV specific responses at baseline and after 12 months
Change in lipodystrophy clinical score and quality of life during the follow-up
Criteria to resume antiretroviral treatment: CD4T cell count below or equal to 300/mm3
The occurrence of an AIDS defining event

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Piketti, MD, Principal Investigator — Hopital Georges Pompidou Paris France; Dominique Costagliola, Study Chair — Inserm U720
Locations (1):
- Service d'immunologie Clinique, Höpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Weiss L, Piketty C, Assoumou L, Didier C, Caccavelli L, Donkova-Petrini V, Levy Y, Girard PM, Burgard M, Viard JP, Rouzioux C, Costagliola D; ANRS 116 SALTO study group. Relationship between regulatory T cells and immune activation in human immunodeficiency virus-infected patients interrupting antiretroviral therapy. PLoS One. 2010 Jul 21;5(7):e11659. doi: 10.1371/journal.pone.0011659. PMID 20657770